CLINICAL TRIAL: NCT01800981
Title: Functionality Assessments in Patients (Adults and Children) Following Treatment With Debrase Compared to Standard of Care (SOC) Protocol MW2012-12-12
Brief Title: Functionality Assessments in Patients (Adults and Children) Following Treatment With Debrase Compared to Standard of Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MW2012-12-12
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Burns, Upper Extremity; Burns, Lower Extremity
Keywords: Functionality; extremities; ROM; Upper and lower Extremity for burned patients
MeSH Terms: conditions — Burns

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Debrase: Patients previously treated with Debrase for burn debridement
- Standard of Care: Patients previously treated with local Standard of Care for burn debridement

SUMMARY:
Once the victim survived the acute phase, the outcome of wound healing, the scarring, became a major medical issue with complications that may lead to cosmetic and functional sequelae. Scar tissue is clinically distinguished from normal skin by an aberrant color, rough surface texture, increased thickness (hypertrophy), contraction, firmness and sometimes, decrease function.

Thus, functional and cosmetic outcomes became at least important as wound closure in assessing wound healing products

DETAILED DESCRIPTION:
This is a multi-center, assessor-blinded study aiming to evaluate the long term functionality in adults and children who have participated in study MW2004-11-02 (previous phase 3 study).

We had previously shown that by using the MVSS scale which includes objective assessment of the physical characteristics of size, shape, volume, color, texture, and pliability as well as structural, mechanical and physiologic characteristics, lower (favorable) scores in Debrase vs. SOC group were observed in sub-groups of highly functional body parts of the hands and feet. This study will include specific functionality evaluation using the "Lower Extremity Functional Scale" test for burns in the lower extremities and the "QuickDASH" outcome measure for burns in the upper extremities as well as range of motion measurements of the joints (knee, ankle, shoulder, elbow and wrist, as relevant).

ELIGIBILITY:
Inclusion Criteria:

* Adults and children who had participated and completed study MW2004-11-02. Patients must be able to sign and dated written informed consent prior to study entry (by Patient or by a guardian, when applicable).

Exclusion Criteria:

* None

Ages: 10 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adults and children who had participated and completed study MW2004-11-02 (previous phase 3 study) will be contacted. Patients who will agree to participate in the study will be invited to the clinic for a one day visit for assessments.
Sampling Method: Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Functionality evaluation using self reported questionnaires and ROM measurements | 2-5 years following to acute treatment
  Functionality evaluation of wounds that have been treated by Debrase or SOC during the previous phase 3 study by:
  1. Self-report questionnaires designed to measure physical function: the "Lower Extremity Functional Scale" test for burns in the lower extremities and the "QuickDASH" outcome measure for burns in the upper extremities.
  2. Range of motion measurements of the following injured joints: knee, ankle, shoulder, elbow, wrist palm and fingers, as relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Koller, PhD, Principal Investigator — Department Head of Burs and Reconstructive Surgery
Locations (1):
- Clinic of Burns and reconstructive surgery hospital, Košice, Slovakia